CLINICAL TRIAL: NCT06839235
Title: A Phase 1/2 Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of ABO-101 in Participants With Primary Hyperoxaluria Type 1 (PH1)
Brief Title: Phase 1/2 Study of ABO-101 in Primary Hyperoxaluria Type 1 (redePHine)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arbor Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABO-101-101
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Primary Hyperoxaluria Type 1 (PH1)
Keywords: PH1; Primary hyperoxaluria; AGXT; CRISPR; Gene Editing; Pharmacokinetics; Pharmacodynamics; ABO-101; redePHine
MeSH Terms: conditions — Primary hyperoxaluria type 1; Hyperoxaluria, Primary

STUDY DESIGN:
Intervention Model Description: Single ascending dose escalation/adaptive design, followed by single dose expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: Part A: Single Ascending Dose Escalation/Adaptive Design (Experimental)
  Interventions: Drug: ABO-101
- Experimental: Part B: Single Dose Expansion (Experimental)
  Interventions: Drug: ABO-101

INTERVENTIONS:
Drug: ABO-101 — Intravenous (IV) infusion

SUMMARY:
The goal of the redePHine study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of ABO-101 in participants with primary hyperoxaluria type 1 (PH1). The trial will consist of 2 Study Periods. During the first Study Period, there will be 2 parts. In Part A, adult participants will be treated with a single ascending dose to identify a recommended dose. In Part B, pediatric participants will be treated with the recommended dose. Following the first Study Period, participants will start Study Period 2, a long-term monitoring program to comply with local and national requirements.

ELIGIBILITY:
Key Inclusion Criteria for Parts A and B

* Documentation of PH1 as determined by genetic analysis confirming pathogenic mutations in the alanine-glyoxylate aminotransferase (AGXT) gene (valid historical laboratory data will be reviewed and approved by the Sponsor)
* Age at time of signing the informed consent/assent form:

  * Part A: ≥18 years to ≤64 years
  * Part B: ≥6 years to <18 years
* 24-hour UOx ≥0.7 mmol/24 hours/1.73 m²
* eGFR ≥30 mL/min/1.73m²
* Weight ≤90 kg

Key Exclusion Criteria for Parts A and B

* Confirmed diagnosis of primary hyperoxaluria type 2 or type 3
* History of a liver, kidney or combined liver/kidney transplant
* Currently on dialysis
* Participant has previously used (within past 24 months) or is currently receiving an approved or investigational urinary oxalate lowering RNA interference (RNAi) or siRNA therapy
* Female participants who are pregnant or breastfeeding (or are planning either during the first 12 months)

Ages: 6 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2043-02 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs), including ABO-101-related TEAEs and serious adverse events (SAEs) | Up to 6 months

SECONDARY OUTCOMES:
Percent change in 24-hour urinary oxalate excretion (UOx) from Baseline to Month 6 | Up to 6 months
Absolute change in UOx corrected for body surface area | Up to 6 months
Percent change in plasma glycolate from Baseline to Month 6 | Up to 6 months
Changes in estimated glomerular filtration rate (eGFR) from Baseline to Month 12 and Month 24 | Up to 24 months
Plasma concentrations for LNP lipids, Cas12i2 mRNA, and guide RNA (gRNA) | Up to 6 months
Urine concentrations for LNP lipids | Up to 6 months
Antidrug antibodies to ABO-101 and anti-Cas protein antibodies | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Winston Yan, MD, PhD, Study Director — Arbor Biotechnologies
Locations (7):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Nucleus Network, Saint Paul, Minnesota
- Hospices Civils de Lyon- Hôpital Femmes Mères Enfants, Lyon, France
- Kindernierenzentrum Bonn, Bonn, Germany
- Heidi Chaker, Sfax, Tunisia
- United Kingdom (2):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided